CLINICAL TRIAL: NCT03921619
Title: Impact of Sling Use on Functional Mobility in a Geriatric Population
Brief Title: Sling Use and Functional Mobility in a Geriatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Assistant Professor, Orthopaedic Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-300002264
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Participants will be asked to perform two balance assessments (Tinetti Balance Scale, Get Up and Go Test) while: 1) not wearing a sling; and 2) wearing a sling on the dominant arm. Additional data will be collected regarding patient frailty with the Edmonton Frail Scale, as well as data regarding sling use and falls in the form of a questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Sling (No Intervention): Participants will perform the balance tests without any added equipment.
- Sling (Dominant) (Experimental): Participants will perform the balance tests with a sling on the dominant arm.
  Interventions: Device: Shoulder Sling

INTERVENTIONS:
Device: Shoulder Sling — soft shoulder sling that is placed around the forearm, with a strap draped over the shoulder
  Arms: Sling (Dominant)

SUMMARY:
Shoulder slings are commonly worn after shoulder surgery. In geriatric patients, painstaking care is taken to reduce any factors that may increase the chance of experiencing a fall. Currently, it is not understood if wearing a sling affects someone's general gait and balance.

DETAILED DESCRIPTION:
Following many shoulder operations, patients are immobilized in an bulky sling with non-weight bearing restrictions for periods of up to 6 weeks. This is necessary to allow for soft tissue healing particularly following repair of rotator cuff tears and shoulder replacement surgeries, two common procedures performed in the elderly population. Previous studies have shown that natural arm swing plays an essential role in maintaining balance and normal gait patterns. Decreased functional mobility and gait impairment has been shown to increase the risk of falls, mortality, and morbidity in an elderly population. However, following upper extremity surgery requiring the use of a sling, targeted therapy for gait and balance training is rarely prescribed. Consequently, the investigators wish to assess whether or not sling use impacts functional mobility test scores in an elderly population. The aim of this project is to maximize perioperative functionality in these patients in efforts to prevent any unanticipated secondary injury.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years of age

Exclusion Criteria:

* Younger than 65 years of age
* Pre-existing cognitive impairment
* Pre-existing mobility impairment
* Pre-existing symptomatic upper or lower extremity disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Tinetti Test | 30 seconds
  Performance-oriented mobility assessment: Components are balance & gait. Patient will be seated in a hard, armless chair and be assessed for balance with all of the following: sitting balance, rising from chair, attempting to rise, immediate standing balance (first 5 sec), standing balance, balance while being nudged, balance with eyes closed, turning 360 degrees, and sitting down. Scored out of 16. The gait portion assesses hesitancy, step length & height, foot clearance, step symmetry, step continuity, path, trunk, and walking time. Scored out of 12. Total score out of 28.
  If score is ≤18, risk of falls is high. If score is 19-23, risk of falls is moderate. If score is ≥24, risk of falls is low.
Timed Up & Go Test | 30 seconds
  Timed stand, walk, and sit test to assess mobility
Edmonton Frail Scale | 1 minute
  Global assessment of patient vulnerability: Domains to be assessed are cognition (clock drawing), general health status (hospitalizations in last year & describing own health), functional independence (how many ADL's require help), social support, medication use (5 or more on a regular basis, adherence to regimen), nutrition (weight loss), mood, continence, and functional performance (timed rising from chair and walking). Scored out of 17, higher scores associated with higher frailty.
  Scoring : 0 - 5 = Not Frail; 6 - 7 = Vulnerable; 8 - 9 = Mild Frailty; 10-11 = Moderate Frailty; 12-17 = Severe Frailty;
Sling / Fall Questionnaire | 1 minute
  General questions about sling use and experiencing a fall. There is no scale associated with this questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No